CLINICAL TRIAL: NCT02647723
Title: Improving Maternal and Child Health Through Prenatal Fatty Acid Supplementation: A Randomized Controlled Study in African American Women Living in Low-income Urban Environments
Brief Title: Improving Maternal and Child Health Through Prenatal Fatty Acid Supplementation
Acronym: NAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB15-0392; R01HD084586 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2024-07-25 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; Child Development
Keywords: Omega-3; Fatty acid; docosahexaenoic; Pregnant; neurodevelopment; stress; urban; african-american; supplement; nutrition; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Docosahexaenoic Acids; Sugars; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral supplement for pregnant women (Experimental): 450 mg/daily of DHA beginning at 10-16 weeks of gestation through the end of pregnancy
  Interventions: Dietary Supplement: DHA
- Sugar pill (Placebo Comparator): 450 mg/daily of sugar pill beginning at 10-16 weeks of gestation through the end of pregnancy
  Interventions: Dietary Supplement: Sugar pill

INTERVENTIONS:
Dietary Supplement: DHA — 2 dietary supplement gel capsules providing 450 mg of DHA twice daily by oral intake for 24 weeks
  Other Names: Omega-3; docosahexaenoic acid
  Arms: Oral supplement for pregnant women
Dietary Supplement: Sugar pill — 2 dietary supplement gel capsules providing 450 mg of soybean oil twice daily by oral intake for 24 weeks
  Other Names: soybean oil
  Arms: Sugar pill

SUMMARY:
The purpose of the study is to test whether nutritional supplementation during pregnancy is associated with 1) improved maternal health during pregnancy; 2) improved infant birth and neurodevelopmental outcomes, and 3) whether the association between nutritional supplementation during pregnancy and infant outcomes is partially mediated by reductions in maternal perceived stress and stress reactivity during pregnancy.

DETAILED DESCRIPTION:
Low-income pregnant women often experience chronic stress and consequently higher levels of stress hormones. In utero exposure to high levels of stress hormones can negatively affect the developing fetus and the infant's capacity for emotion and behavioral regulation. This program of research is designed to reduce the negative impact of prenatal stress on infant health and development via nutritional supplementation of docosahexaenoic acid (DHA) during pregnancy. DHA is a long-chain polyunsaturated fatty acid member of the omega-3 fatty acid family. DHA is found in its highest concentrations in neural cell membranes, affecting receptor function, neurotransmitter uptake, and signal transmission. There is growing evidence that low levels of dietary DHA intake are associated with suboptimal response to stress and that DHA supplementation can modulate stress response.

One hundred sixty-two pregnant women will be randomly assigned to receive 450 mg/daily of DHA or placebo beginning at 9-12 weeks of gestation through the end of pregnancy. Perceived stress, stressful life events, anxiety, and depression, inflammatory markers, DHA levels and response to a laboratory stressor will be assessed at baseline and at 24, 30, and 36 weeks of pregnancy. Neonatal outcomes (e.g., gestational age, birth weight, delivery complications) will be collected from medical records, and infant neurodevelopmental outcomes and stress reactivity will be assessed at 1, 4 and 9 months of age. Coded data will be analyzed by the Investigators at University of Chicago and University of Pittsburgh

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 34
* Household recipient of public assistance (e.g. Medicaid insurance) due to low income
* Low levels of DHA consumption as defined as less than two fish servings per week

Exclusion Criteria:

* Reports of known medial complications
* Regular use of steroid medications, alcohol, cigarettes, or illegal substances (by maternal report)
* Use of blood thinners or anti-coagulants
* Use of psychotropic medications
* Allergy to iodine and/or soy

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Keenan, Ph.D, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Active recruitment from the University of Chicago Medical Center and affiliated Federally Qualified Health Centers (FQHC) occurred between 2016 and 2021.
Period: Overall Study
Arm/Group | Oral Supplement for Pregnant Women | Sugar Pill
Started | 112 | 56
Completed | 112 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Supplement for Pregnant Women | Sugar Pill | Total
Number analyzed (Participants) | 112 | 56 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 56 | 168
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.80 (4.27) | 25.47 (4.11) | 25.69 (4.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 56 | 168
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 112 | 56 | 168
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 112 | 56 | 168

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Perceived Stress Scale (PSS) Score From Visit 1 to Visit 4
Description: Will be assessed at baseline and at 24, 30, and 36 weeks of pregnancy, and at 1, 4 and 9 months after giving birth.
  The Perceived Stress Scale score is obtained by summing the points awarded to the 10 items and it ranges from 0 to 40 where:
  0-13 - Low stress 14-26 - Moderate stress 27-40 - High perceived stress
Time Frame: 16 months
Population: Of the 168 participants recruited, 127 had PSS data for all 4 visits.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Oral Supplement for Pregnant Women | Sugar Pill
Number analyzed (Participants) | 86 | 41
change in score on a scale | 2.33 (6.81) | 3.65 (6.66)

2. Primary Outcome: Average Change in Perceived Stress Scale (PSS) Score From Visit 1 to Visit 3
Description: as for outcome 1
Time Frame: 12 months
Population: Of the 168 participants recruited, 133 had PSS data for visits 1, 2 and 3.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Oral Supplement for Pregnant Women | Sugar Pill
Number analyzed (Participants) | 92 | 41
change in score on a scale | 1.91 (6.09) | 3.56 (7.49)

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | Oral Supplement for Pregnant Women | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/56
Other Adverse Events (participants affected / at risk) | 0/112 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT02647723/Prot_SAP_000.pdf